CLINICAL TRIAL: NCT01474421
Title: A Multi-centre, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multiple Oral Dose Study to Assess the Efficacy, Safety and Tolerability of AQW051 in Reducing L-dopa Induced Dyskinesias in Parkinson's Patients With Moderate to Severe L-dopa Induced Dyskinesias
Brief Title: Safety and Efficacy of AQW051 in L-dopa Induced Dyskinesias in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAQW051A2209; 2011-001092-39 (EudraCT Number)
Record Dates: First submitted 2011-10-05; First posted 2011-11-18 (Estimated); Last update posted 2020-12-24 (Actual); Status verified 2017-05

CONDITIONS: Dyskinesias; Drug-induced
Keywords: Parkinson's disease; Dyskinesia; Movement disorders; L-dopa
MeSH Terms: conditions — Dyskinesias; Parkinson Disease; Movement Disorders | interventions — 3-(6-p-tolylpyridin-3-yloxy)-1-azabicyclo(2.2.2)octane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AQW051 High Dose (Experimental): AQW051 high dose daily given orally for 28 days.
  Interventions: Drug: AQW051
- AQW051 Low Dose (Experimental): AQW051 low dose daily given orally for 28 days.
  Interventions: Drug: AQW051
- Placebo (Placebo Comparator): Placebo daily given orally for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AQW051 — Patients will receive AQW051 in a high dose once daily orally for 28 days.
  Arms: AQW051 High Dose
Drug: AQW051 — Patients will receive AQW051 in a low dose once daily orally for 28 days.
  Arms: AQW051 Low Dose
Drug: Placebo — Patients will receive placebo once daily orally for 28 days.
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability and efficacy of AQW051 in treating moderate to severe L-dopa induced dyskinesias (movement disorders) in patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease
* Patients with dyskinesias for at least 3 months
* Patients with moderate to severe dyskinesias
* Patients on L-dopa treatment for at least 3 years

Exclusion Criteria:

* Patients with atypical Parkinson's disease
* Patients who have had prior surgery for Parkinson's disease
* Patients who are cognitively impaired, have psychosis, have confusional states or hallucinate
* Patients who received neuroleptics or anti-psychotics within 2 months
* Women of child-bearing potential

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2011-09-15 (Actual); Primary Completion 2013-02-21 (Actual); Study Completion 2013-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Modified Abnormal Involuntary Movement Scale (mAIMS)score | Baseline, Day 28
  Dyskinesia with a maximal score of 24.
Change in Unified Parkinson's Disease Rating Scale (UPDRS) - Part III score | Baseline, Day 28
  Anti-parkinsonian effect in PD patients.
Safety and tolerability | Up to Day 42
  Safety and tolerability of AQW051 as measured by the number of participants with adverse events, any clinically significant abnormalities in safety labs or electrocardiograms (ECGs), and relevant orthostatic changes in blood pressure

SECONDARY OUTCOMES:
Lang-Fahn Activities of Daily Living Dyskinesia Scale (LFADLDS) | Up to Day 42
  Assesses the degree to which dyskinesia interferes with five activities of daily living, with a higher score indicating more severe impairment.
Unified Parkinson's Disease Rating Scale (UPDRS) - Part IV, #32-33 | Up to Day 42
  Dyskinesias as a percentage of the day, and disability due to dyskinesia during the previous week.
Track-PD | Up to Day 42
  Objective measures of motor function.
CogState | Up to Day 28
  Cognitive function, including simple and choice reaction time, episodic visual and verbal memory, working memory, planning and strategy, and executive function.
Area under the curve (AUC[0-24hr]) of AQW051 | Day 28

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (24):
- United States (4):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, Manhasset, New York
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Cleveland, Ohio
- France (11):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Clermont Fd
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (8):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Gera
  - Novartis Investigative Site, Haag
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Roma, RM, Italy

REFERENCES:
- [Result] Trenkwalder C, Berg D, Rascol O, Eggert K, Ceballos-Baumann A, Corvol JC, Storch A, Zhang L, Azulay JP, Broussolle E, Defebvre L, Geny C, Gostkowski M, Stocchi F, Tranchant C, Derkinderen P, Durif F, Espay AJ, Feigin A, Houeto JL, Schwarz J, Di Paolo T, Feuerbach D, Hockey HU, Jaeger J, Jakab A, Johns D, Linazasoro G, Maruff P, Rozenberg I, Sovago J, Weiss M, Gomez-Mancilla B. A Placebo-Controlled Trial of AQW051 in Patients With Moderate to Severe Levodopa-Induced Dyskinesia. Mov Disord. 2016 Jul;31(7):1049-54. doi: 10.1002/mds.26569. Epub 2016 Mar 15. PMID 26990766
- See also: Results for CAQW051A2209 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=10163